CLINICAL TRIAL: NCT04799561
Title: Virtual Prehabilitation of Surgical Cancer Patients in Times of the Covid-19 Pandemic
Brief Title: Teleprehabilitation for Surgical Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Montreal General Hospital (Other); Peri Operative Program, Montreal (Unknown)
Responsible Party: Principal Investigator, Franco Carli, Principal Investigator and Professor of Anesthesia, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MUHC-2021-6730
Record Dates: First submitted 2021-03-01; First posted 2021-03-16 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Abdominal Cancer; Thoracic Cancer
Keywords: Telehealth; Telemedecine; Prehabilitation; Supportive Care

STUDY DESIGN:
Intervention Model Description: This QI study will include one group of 100 patients who will receive distance-delivered support for all components of the home-based prehabilitation regimen in addition to 2 months of follow-up post-surgery. The program will include: exercise, nutrition, mental well-being and, if needed, smoking cessation. The technologies (a tablet and an active lifestyle watch) will be used to provide counselling, educate patients on lifestyle modifications and assess adherence remotely. Telephone calls will also be made on a weekly basis, if participants were unable to attend their video-conferencing counselling sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Teleprehabilitation cohort (Experimental): Patients in this single-arm study will receive multimodal teleprehabilitation.
  Interventions: Behavioral: Multimodal Teleprehabilitation

INTERVENTIONS:
Behavioral: Multimodal Teleprehabilitation — Exercise Prescription: patients will be instructed on how to perform aerobic exercise (5 times/week: minimum 30-minute/day) and resistance training (3 times/week: 2-3 sets of 6-8 exercises repeated 8-12 times) at home. Exercise counseling will be weekly, using the video-conferencing application (Zoom).
  Nutrition: nutritional status and dietary intake will initially be assessed by the nutritionist using zoom. All patients will receive daily whey protein supplements. Special precautions will be considered if patients have specific medical conditions.
  Psychosocial intervention: Patients will have access to 1.5 hours of mental relaxation and coping mechanisms session within the first week of enrolment, using Zoom.
  Smoking Cessation: Patients with smoking habits will meet with a respiratory specialist using Zoom, who will establish recommendations and contact the physician for the recommended smoking cessation protocol.
  More counseling sessions will be provided as needed.
  Other Names: Virtual Prehabilitation

SUMMARY:
There is a general concern that the backlog of cancer patients waiting for surgery during this period is going to increase and the general impact on patients isolated in their homes is going to cause potential physiological and psychological impairments. Therefore, we propose a distanced-delivered personalized home-based prehabilitation program to all cancer patients scheduled for surgery at the MUHC. The program will be delivered by qualified professionals, supported by technology provided by POP, to all cancer patients waiting for surgery, addressing the patients' risk factors in patients' pandemic reality perspective. Participant contacts will primarily occur virtually using technologies such as video conferencing and digital applications. This will enable us to continue to support people with cancer and deliver safe remote counseling by specialist healthcare providers in their own homes, whilst adhering to the Governmental guidelines on social distancing, self-isolation and shielding.

DETAILED DESCRIPTION:
The current project aims to improve the quality of care delivered to oncologic surgical candidates during the COVID-19 pandemic. The specific objectives of the study are: 1. to assess the feasibility of a distance-delivered prehabilitation program to oncologic surgical candidates in light of the current global pandemic, 2. to measure the effect of technology-supported prehabilitation on preoperative and postoperative functional capacity and clinical outcomes, and 3. To qualitatively investigate the impact of distance-delivery of prehabilitation on health-related quality of life, anxiety and depression, which may be exacerbated by the current global phenomenon.

To do so, a convenient study group of 100 patients on the waiting lists to undergo elective thoracic and abdominal surgery, initially at the Montreal General Hospital (MGH) will be recruited over the next year and a half.

Program:

The program for the current study will consist of two parts, the first being individual counseling with different healthcare professionals, the second component would be a home-based prehabilitation program for patients awaiting their surgery. The healthcare providers available for participants' respective needs include exercise physiologist (a), nutritionists (b), psychosocial (c), and if needed smoking cessation (d) personnel who would contact patients via phone, and a videoconferencing platform (Zoom) if possible, facilitated by the use of the tablet.

Exercise physiologists will follow-up with patients regularly throughout the continuum of care (before and after their surgery) and refer them to the relevant specialists as needed.

The patients will also have access to premade videos prepared by POP to provide additional support in their application of the preoperative recommendations: physical activity (aerobic, resistance, and flexibility), nutrition optimization (healthy eating, improving protein and energy intake, portion size, glycemic control), psychological exercises (breathing exercise, relaxation, imaging, visualization) and smoking cessations. These videos will be available to the patients on their tablets, in addition, the exercises will be demonstrated in the booklets.

Outcome Measures:

All outcomes will be captured via patient chart review, self-report questionnaires, data collected from the Polar watch, and digital surveys. Chart review outcomes include the length of hospital stay, surgical and postoperative complications.

The primary outcome of the current study is to assess the feasibility of distance-delivery of Prehabilitation to these high-priority cancer patients using a digital platform. In order to ascertain if the program was feasible, the evaluation criteria included quantitative measures such as recruitment rate, adherence to program (self-reported measures and crude data from the polar), program completion rate, frequency of technological failures, adverse events, in addition to qualitative measures such as rationale for refusal to participate, low compliance and drop-outs.

Secondary outcomes also include parameters of functional health, nutritional and metabolic status, self-reported outcomes, and surgical outcomes.

Potential confounding variables:

The current study will investigate a diverse patient population. A large degree of variability is to be expected in the observed functional and clinical outcomes. Several factors are known to affect patient prognosis and recovery, among them baseline BMI, smoking status, comorbidities (CCI), type of cancer, neoadjuvant therapies (type and duration) and duration of the prehabilitation program. Therefore, the current study will investigate the impact each factor on the reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults scheduled for elective cancer surgery that is delayed due to COVID-19 referred by a surgeon;
* Covered by the RAMQ
* Have medical clearance to exercise (as provided on the physician referral);
* Are able to understand English or French.

Exclusion Criteria:

* N.A.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-03-12 (Actual); Primary Completion 2022-09-15 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | Through study completion, for an expected duration of of 1.5 year.
  Recruitment rate is defined as the number of participant recruited, compared to the number of eligible participant contacted.
Adherence | Through study completion, for an expected duration of of 1.5 year.
  based on self-reported measures and data from the polar watch, compared to prescribed intervention
Program Completion Rate | Through study completion, for an expected duration of of 1.5 year.
  The completion rate is defined as the number of participant completing all evaluations, compared to the number of participants recruited.
frequency of Technological Failures | Through study completion, for an expected duration of of 1.5 year.
  Frequency of technological failures is defined as the number of any technological challenge that would prevent participants from doing their interventions or contacting the research team member.
Intervention-Related Adverse Events | Through study completion, for an expected duration of of 1.5 year.
  Intervention-related adverse events is defined as any event that would cause harm to patients' physical or mental health.
Rational for Refusal to Participate | Through study completion, for an expected duration of of 1.5 year.
  When possible, patients' rational for refusing to participate in the project was collected.
Rational for Low Compliance | Through study completion, for an expected duration of of 1.5 year.
  When possible, participant's rational for low compliance to the project was collected.
Rational for Drop-Outs | Through study completion, for an expected duration of of 1.5 year.
  When possible, participant's rational for abandoning the project was collected.

SECONDARY OUTCOMES:
30 Second Sit-to-Stand | During baseline assessment (beginning of prehabilitation period; T0), at the preoperative assessment (within the 24 hours prior to surgery; T1) and further at the 4- (T2) and 8-weeks (T3) follow-ups after surgery
  Assessed the strength of the lower body, by sitting on a chair and standing up as many times as possible during 30 seconds.
Time-Up and Go (TUG) | During baseline assessment (beginning of prehabilitation period; T0), at the preoperative assessment (within the 24 hours prior to surgery; T1) and further at the 4- (T2) and 8-weeks (T3) follow-ups after surgery
  Assessed mobility, balance and locomotor performance associated to the tasks of walking and turning. The patients starts seated, and needs to stand up, walk turn around a cone and sit back down as fast as possible, the results is the numbers of seconds to perform the 3-meter distance to a cone and back.
2- or 6-Minute Walk Test | During baseline assessment (beginning of prehabilitation period; T0), at the preoperative assessment (within the 24 hours prior to surgery; T1) and further at the 4- (T2) and 8-weeks (T3) follow-ups after surgery
  The 2- or 6-minute walk test is a functional capacity measure, surrogate to the assessment of cardiopulmonary capacities. The patient walks in a 20-meter corridor, back and forth, for 2 or 6 minutes and the result of the test is the distances traveled in meters.
Abridged-Scored Patient-Generated Subjective Global Assessment (PG-SGA) | During baseline assessment (beginning of prehabilitation period; T0), at the preoperative assessment (within the 24 hours prior to surgery; T1) and further at the 4- (T2) and 8-weeks (T3) follow-ups after surgery
  Assessed the state of nutrition, classification A, B or C ( B and C being states of nutritional risk).
Body Mass Index (BMI) | During baseline assessment (beginning of prehabilitation period; T0), at the preoperative assessment (within the 24 hours prior to surgery; T1) and further at the 4- (T2) and 8-weeks (T3) follow-ups after surgery
  Assessed the body composition, ranging 18 to 30 (>30 is obesity, and <18 is malnourished).
CRP | During baseline assessment (beginning of prehabilitation period; T0)
  Assessed the degree of inflammation (>10mg/L indicates high inflammation )
Serum Albumin | During baseline assessment (beginning of prehabilitation period; T0)
  Assessed the degree of inflammation (<35g/L indicates high inflammation)
Duke Activity Status Index (DASI) | During baseline assessment (beginning of prehabilitation period; T0), at the preoperative assessment (within the 24 hours prior to surgery; T1) and further at the 4- (T2) and 8-weeks (T3) follow-ups after surgery
  Assessed the level of physical activity and is measured in 12 questions, going up to a score of 58 (58 being the best score).
Quality of Life (EQ5D) | During baseline assessment (beginning of prehabilitation period; T0), at the preoperative assessment (within the 24 hours prior to surgery; T1) and further at the 4- (T2) and 8-weeks (T3) follow-ups after surgery
  Assessed the quality of life of the previous week, on a scale of 0 to 100 ( 100 being the best health).
The Hospital Anxiety and Depression Scale (HADS) | During baseline assessment (beginning of prehabilitation period; T0), at the preoperative assessment (within the 24 hours prior to surgery; T1) and further at the 4- (T2) and 8-weeks (T3) follow-ups after surgery
  Assessed the degree of anxiety and depression, separately, ranging from 0 to 18 respectively (18 being the worst score).
Distress Thermometer | During baseline assessment (beginning of prehabilitation period; T0), at the preoperative assessment (within the 24 hours prior to surgery; T1) and further at the 4- (T2) and 8-weeks (T3) follow-ups after surgery
  Assessment of the level of anxiety and distress, on a scale from 0 to 10 (10 being the worst score).
The WHO Disability Assessment Schedule v2.0 (WHODAS) | During baseline assessment (beginning of prehabilitation period; T0), at the preoperative assessment (within the 24 hours prior to surgery; T1) and further at the 4- (T2) and 8-weeks (T3) follow-ups after surgery
  the WHO Disability Assessment Schedule is a scale of disability free survival, measured at different times,
The Energy Expenditure (CHAMPS) | During baseline assessment (beginning of prehabilitation period; T0), at the preoperative assessment (within the 24 hours prior to surgery; T1) and further at the 4- (T2) and 8-weeks (T3) follow-ups after surgery
  the energy expenditure related to physical activities of daily living, measured in kilocalories/kg/week.
The Clavien-Dindo Classifications(CDC) | During the post-operative period, data collected on average up to 2 months after the surgery date.
  The Clavien-Dindo Classifications(CDC) indicates the resource utilization of complication post-operatively, ranging from 0 to 4 (4 being patient admitted to the intensive care).
The Comprehensive Complication Index (CCI) | During the post-operative period, data collected on average up to 2 months after the surgery date.
  The comprehensive complication index (CCI) is a score of the r severity of post-operative complications, ranging from 0 to 100 (100 being mortality).
The 30-day Mortality | During the post-operative period, for a month after the surgery date.
  The 30-day mortality will assess the number of deaths within the first 30 days post-surgery.
Length of Intensive Care Stay | During the post-operative period, data collected on average up to 2 months after the surgery date.
  Length of intensive care stay will be assessed as the number of hours from arrival to the unit.
Days with a chest tube | During the post-operative period, data collected on average up to 2 months after the surgery date.
  Days with a chest tube will be assessed as the number of days and hours for the last day, if applicable.
Length of Hospital Stay | During the post-operative period, data collected on average up to 2 months after the surgery date.
  Length of Hospital Stay will be assessed as a number of post-operative hours until discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Muhc-Rimuhc, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lambert G, Drummond K, Tahasildar B, Carli F. Virtual Prehabilitation in Patients With Cancer Undergoing Surgery During the COVID-19 Pandemic: Protocol for a Prospective Feasibility Study. JMIR Res Protoc. 2022 May 6;11(5):e29936. doi: 10.2196/29936. PMID 35522464

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-05): https://cdn.clinicaltrials.gov/large-docs/61/NCT04799561/Prot_SAP_000.pdf